CLINICAL TRIAL: NCT07277153
Title: Clinical Study on the Effect of Tegileridine on Postoperative Pain in PatientsUndergoing Abdominal Surgery：A Randomized Controlled Double-blind Trial.
Brief Title: Clinical Study on the Effect of Tegileridine on Postoperative Pain in Patients Undergoing Abdominal Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xin Chen (Other)
Collaborators: The Second Affiliated Hospital of Hainan Medical University (Other)
Responsible Party: Sponsor-Investigator, Xin Chen, Associate Researcher,the Second Affiliated Hospital of Hainan Medical University, Hainan Medical College
Organization: Hainan Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HNMU2H-POPABD-CN-2025; No.823RC592 (Other: Hainan Provincial Natural Science Foundation of China)
Record Dates: First submitted 2025-11-27; First posted 2025-12-11 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Laparoscopic Surgery for Cholecystitis
Keywords: Tegileridine; Abdominal surgery; Postoperative pain; Moderate-to-severe pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution; Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pre-incision tegileridine (T1 group） (Experimental): Tegileridine 1 mg IV, diluted to 10 mL in 0.9% sodium chloride, infused over 10 minutes after anesthesia induction and before skin incision.
  At skin closure, a matched 10 mL normal saline infusion is given. Rescue analgesia is permitted per institutional practice.
  Interventions: Drug: Tegileridine (tegileridine fumarate injection, IV)
- End-of-surgery tegileridine（T2 group） (Experimental): After anesthesia induction and before skin incision, a matched 10 mL normal saline infusion is given.
  At skin closure, tegileridine 1 mg IV, diluted to 10 mL in 0.9% sodium chloride, is infused over 10 minutes. Rescue analgesia is permitted per institutional practice.
  Interventions: Drug: Tegileridine (tegileridine fumarate injection, IV)
- Placebo Comparator（C group） (Placebo Comparator): 0.9% sodium chloride (normal saline, IV) - matched 10 mL infusion over 10 minutes administered at the alternate timepoint to maintain blinding.
  Interventions: Other: 0.9% Normal Saline (0.9% Sodium Chloride) injection

INTERVENTIONS:
Drug: Tegileridine (tegileridine fumarate injection, IV) — Tegileridine (tegileridine fumarate injection, IV) is a small-molecule μ-opioid receptor agonist with G-protein-biased signaling (relative to β-arrestin-2 recruitment), developed by Jiangsu Hengrui for postoperative analgesia. It is administered intravenously and was first approved in China in January 2024 for the treatment of moderate-to-severe pain after abdominal surgery; in this study, tegileridine is used as part of standardized multimodal analgesia according to protocol. In China it is regulated as a narcotic drug.
  Arms: End-of-surgery tegileridine（T2 group）; Pre-incision tegileridine (T1 group）
Other: 0.9% Normal Saline (0.9% Sodium Chloride) injection — 0.9% sodium chloride (normal saline, IV) - matched 10 mL infusion over 10 minutes administered at the alternate timepoint to maintain blinding.
  Arms: Placebo Comparator（C group）

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of tegileridine fumarate injection for postoperative analgesia in adults experiencing moderate-to-severe pain after abdominal surgery. Participants will be randomized to receive intravenous tegileridine or matching placebo as part of a standardized multimodal analgesia protocol; all patients will have access to rescue opioid analgesia per institutional practice. The primary objective is to determine whether tegileridine improves postoperative pain control during the first 24-48 hours after surgery. Secondary objectives include comparing cumulative opioid consumption, time to first rescue analgesia, patient-reported satisfaction with pain control, recovery milestones (e.g., time to ambulation), and the incidence of adverse events such as nausea, vomiting, sedation, respiratory depression, pruritus, and constipation. Safety will be monitored throughout the study with predefined stopping and reporting procedures. The results aim to inform whether tegileridine can provide effective and well-tolerated analgesia for patients with moderate-to-severe postoperative pain following abdominal procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years; BMI 18-35 kg/m²; ASA physical status I-III.

  * Diagnosed with symptomatic gallbladder stone disease and scheduled for elective laparoscopic cholecystectomy under general anesthesia; expected procedure duration ≥60 minutes and postoperative hospitalization ≥24 hours.

    * Investigator expects moderate-to-severe postoperative pain; willing to receive standardized multimodal analgesia and protocolized rescue analgesia.

      * Able to understand pain scales (NRS/VAS) and provide written informed consent.

        * Women of childbearing potential: negative pregnancy test within 72 hours preoperatively and agreement to use effective contraception through 30 days after last dose.

Exclusion Criteria:

* Known hypersensitivity to opioids or any component of the study drug.

  * Chronic opioid use/tolerance (e.g., ≥30 mg MME/day for ≥7 consecutive days within 30 days pre-op) or current methadone/buprenorphine therapy.

    * Planned/required neuraxial analgesia (epidural/spinal), continuous peripheral nerve blocks, or use of long-acting local anesthetic formulations that would confound postoperative pain assessment; brief intraoperative wound infiltration with short-acting local anesthetics is allowed if standardized.

      * Significant respiratory disease (e.g., uncontrolled obstructive sleep apnea, GOLD III-IV COPD) or anticipated postoperative mechanical ventilation >24 hours.

        ⑤Severe hepatic or renal impairment (Child-Pugh B/C; eGFR <30 mL/min/1.73 m²; or ALT/AST >3×ULN with total bilirubin >2×ULN).

        ⑥Clinically unstable cardiovascular or cerebrovascular disease (e.g., shock, uncontrolled arrhythmias, myocardial infarction or stroke within 6 months), or persistent SBP <90 mmHg.

        ⑦Concomitant medications that cannot be safely withheld: MAO inhibitors within 14 days; strong CNS depressants requiring continued use (e.g., benzodiazepines/barbiturates); mixed agonist-antagonist opioids (e.g., nalbuphine, buprenorphine) within 7 days.

        ⑧Severe psychiatric/neurologic disease or communication/cognitive impairment precluding valid pain scoring or follow-up.

        ⑨Pregnancy or breastfeeding; unwillingnebass to use contraception.

        ⑩Substance abuse (alcohol or drugs) within 12 months.

        ⑪Participation in another interventional study with study drug/device within 30 days.

        ⑫Any other condition that, in the opinion of the investigator, makes participation unsafe or impractical (e.g., severe active infection, planned ICU admission).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-10-18 (Actual); Primary Completion 2025-12-14 (Actual); Study Completion 2025-12-14 (Actual)

PRIMARY OUTCOMES:
Postoperative Visual Analog Scale(VAS)Pain Scores at Multiple Time Points | 2 hours ( h), 6 h, 12 h, 24 h, 36 h and 48 h after surgery
  Pain intensity is assessed with the 10-cm Visual Analog Scale (minimum 0 = no pain, maximum 10 = worst imaginable pain) at rest by blinded assessors at 2 h, 6 h, 12 h, 24 h, 36 h and 48 h after surgery; lower scores indicate less pain. When rescue analgesia is required, VAS is recorded immediately before rescue dosing.

SECONDARY OUTCOMES:
Intraoperative opioid consumption | Perioperative (induction of anesthesia to end of surgery).
  Total intraoperative opioid use, expressed in intravenous morphine milligram equivalents.
Quality of Recovery-15 (QoR-15) Score | Day 1 and Day 2 postoperatively.
  Researchers assist patients in completing the QoR-15 questionnaire (minimum 0 = very poor quality of recovery, maximum 150 = excellent quality of recovery); higher scores indicate better quality of recovery.
Richmond Agitation and Sedation Scale(RASS) | Immediately before removal of the endotracheal tube (Postoperative Day 0).
  The research team assigns a RASS score (minimum -5 = unarousable, maximum +4 = combative; scores closer to 0 indicate an alert and calm state) by observing the patient immediately before tracheal extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology,the Second Affiliated Hospital of Hainan Medical University, Haikou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuang Y, Shen L, Luo Y, Li B, Su X, Zhou Z, Zhao Y. Biased mu-opioid receptor agonists for postoperative pain: Balancing efficacy and safety in clinical translation. Pharmacol Res. 2025 Nov;221:107994. doi: 10.1016/j.phrs.2025.107994. Epub 2025 Oct 12. No abstract available. PMID 41086976
- [Result] Huang L, Jiang H, Huang Y, Li J. Exploring Pharmacokinetic interactions between SHR8554, a micro-opioid receptor biased agonist, and Itraconazole in healthy Chinese subjects. Sci Rep. 2025 Jul 2;15(1):22635. doi: 10.1038/s41598-025-98697-3. PMID 40593123
- [Result] Feng Y, Yang G, Zhang P, Li L, Tian J, Wang Y, Chu Q. The Analgesic Effect of Tegileridine in Older Adult Patients After Laparoscopic Abdominal Tumor Surgery: Study Protocol for a Randomized Controlled Trial. Pain Ther. 2026 Feb;15(1):433-441. doi: 10.1007/s40122-025-00798-4. Epub 2025 Nov 20. PMID 41264221
- [Result] Dhillon S. Correction: Tegileridine: First Approval. Drugs. 2024 Aug;84(8):1011. doi: 10.1007/s40265-024-02079-4. Epub 2024 Aug 12. No abstract available. PMID 39133436
- [Result] Kissin I. Preemptive analgesia. Anesthesiology. 2000 Oct;93(4):1138-43. doi: 10.1097/00000542-200010000-00040. No abstract available. PMID 11020772
- [Result] Zhao Y, Lu Z, Song X, Xie H, Xiao X, Wang G, Zhou Q, Zhang Q, Liu L, Lan Z, Bai N, Wang H, Pan Z, Dong L, Lin X, Chen G, Wang Q, Dong J, Deng J, Nan Y, Zhang J, Zhou X, Huang Y, Chen Y, He H, Yang Y, Yao D, Jia J, Jin S, Zhang Y, Luo Z, Li J, Zhang L, Wang F, Jing J, Zhu J, Li L, Wang G, Guo H, Wang Q, Su D, Yu W, Gu X. Efficacy and safety of SHR8554 on postoperative pain in subjects with moderate to severe acute pain following orthopedic surgery: A multicenter, randomized, double-blind, dose-explored, active-controlled, phase II/III clinical trial. Pharmacol Res. 2025 Feb;212:107576. doi: 10.1016/j.phrs.2025.107576. Epub 2025 Jan 3. PMID 39755132